CLINICAL TRIAL: NCT05208801
Title: Analgesic Effect of Intrathecal Morphine Combined With Low Dose Local Anesthetics on Postoperative Analgesia After Liver Resection: A Randomized, Controlled Preliminary Study
Brief Title: Analgesic Effect of Intrathecal Morphine Combined With Low Dose Local Anesthetics on Postoperative Analgesia After Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2018-0838
Record Dates: First submitted 2021-12-15; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Patients Receiving Hepatectomy Under General Anesthesia
MeSH Terms: interventions — Administration, Cutaneous; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): a sham procedure of 2 ml of 1% lidocaine injected percutaneously using the initial 25G needle
  Interventions: Drug: Percutaneous injection
- Morphine (Active Comparator)
  Interventions: Drug: Morphine
- Morphine+bupivicaine (Experimental)
  Interventions: Drug: Morphine+Bupivacaine

INTERVENTIONS:
Drug: Percutaneous injection — A sham procedure of 2 ml of 1% lidocaine injected percutaneously using the initial 25G needle for local anesthetics
  Arms: Control
Drug: Morphine — Intrathecal injection of morphine 400mcg
  Arms: Morphine
Drug: Morphine+Bupivacaine — Intrathecal injection of 5mg of 0.5% bupivacaine chloride
  Arms: Morphine+bupivicaine

SUMMARY:
Efficient postoperative pain control plays a vital part in the management of patients after surgery. In particular, major surgeries including hepatectomy cause intense postoperative pain that may result in cardiovascular or respiratory complications post-surgery. One of the current methods of postoperative pain control after hepatectomy involves a multimodal approach including intrathecal morphine injection immediately prior to surgery. Because morphine alone is inadequate for immediate postoperative pain control due to a late peak effect time of 6 hours, current literature advocates a combination injection including bupivacaine. However, higher doses of bupivacaine may inadvertently cause motor block or hemodynamic side effects. The aim of this study was to compare the effectiveness and side effects of intrathecal morphine combined with low dose bupivacaine against intrathecal morphine alone and no intrathecal injection.

DETAILED DESCRIPTION:
All patients enrolled in the current study will receive intrathecal injections immediately prior to general anesthesia. The patient will be on his or her side in the fetal position and after palpating the back to secure the space between the 3rd and 4th lumbar spine, the area will be properly disinfected and draped with a sterile towel. Using a 25G needle, a small volume of 1% lidocaine will be injected at the proposed puncture site. For the control group, 2ml of 1% lidocaine will be injected subcutaneously with the 25G needle used during local anesthetic injection. For the morphine group and the morphine + bupivacaine group, a 25G pencil point spinal needle will be used to advance into the intrathecal space. After confirming intrathecal position of the needle by CSF regurgitation, morphine 400mg or morphine 400mcg+ bupivacaine 5mg each to a total volume of 2ml will be injected. Afterwards, all patients will undergo general anesthesia by the same method.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years to no upper limit
2. Patients receiving liver resection under general anesthesia (Including open surgery and laparoscopic surgery)
3. American Society of Anesthesiologists (ASA) physical status 1,2

Exclusion Criteria:

1. Patients presenting with coagulopathy prior to surgery
2. Patients with neurological deficits
3. Patients with spinal anomaly or disorders
4. Patients with allergies to opioids or local anesthetics
5. Patients with severe respiratory, cardiovascular, renal, or hepatic disorders
6. Severe systemic infection or infections involving proposed intrathecal injection site
7. Patients with severe psychological disorders severe that may interfere with pain evaluation
8. Patients with chronic diseases that require opioids

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-04-18 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesic | First 72 hours after surgery
  Time to first rescue analgesic during the first 72 hours after surgery (hr) was our primary outcome.

SECONDARY OUTCOMES:
Pain score after surgery (visual analogue scale, VAS) | 30 minutes, 1 hours upon arrival of the Postoperative anesthesia care unit(PACU), 5 hours post surgery, 1 day post-surgery
  Visual analogue scale is a validated subjective measure for acute and chronic pain. Scores are measured on 10cm line where 0 represents no pain to 10cm representing the worst pain.
Total fentanyl dose administered via intravenous patient-controlled analgesia (PCA) | First 48 hour post surgery
  Further assessment of pain control was done by comparing total opioid dosage via PCA.
Additional rescue analgesics given to the patient | until 3 days post-surgery.
  Rescue analgesics were given only upon patients request. This was evaluated for further assessment of pain control.
Sensory and motor block | 30 minutes, 1 hours upon arrival of the Postoperative anesthesia care unit (PACU), 5 hours post surgery, 1 day post-surgery
  Sensory and motor block was assessed for prolonged effects of intrathecal injection.
Presence of complications (headache, nausea/vomiting, pruritus, respiratory depression, somnolence, low blood pressure, tingling, and shivering) | first 3 days post surgery
  Common side effects to morphine or bupivacaine injections were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Nye Koo, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided